CLINICAL TRIAL: NCT05987579
Title: Surgical Treatment of Stage T3 Squamous Cell Carcinomas of the Scalp
Status: Active, not recruiting | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-2706
Record Dates: First submitted 2023-07-20; First posted 2023-08-14 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Squamous Cell Carcinoma; Surgery; Cancer Head Neck
MeSH Terms: conditions — Carcinoma, Squamous Cell; Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study examines tumor- en surgical characteristics of stage T3 cutaneous squamous cell carcinomas on the scalp, diagnosed between 2010 and 2018. Histological data and patient- and tumor characteristics were collected.

DETAILED DESCRIPTION:
Cutaneous squamous cell carcinoma is the second most common type of non-melanoma skin cancer, following basal cell carcinoma. Following the American Joint Committee on Cancer Tumour, Node and Metastasis (TNM) Classification of Malignant Tumors staging system (TNM8), T3 cutaneous squamous cell carcinomas comprise an interesting group, especially on the scalp, because of the thin subcutaneous fat layer. According to the TNM8 criteria, T3 include all cutaneous squamous cel carcinomas with greatest tumor dimension ≥4cm, tumors with minimal bone erosion or perineural growth (defined as involvement of the nerve sheath of a nerve lying deeper than the dermis or measuring 0.1mm or larger in caliber or showing clinical or radiographic involvement of nerves without invasion of the skull base) or with deep invasion. Deep invasion is defined as invasion deeper than the subcutaneous fat or a tumor thickness >6mm. The scalp has a natural anatomical and oncological barrier for extension in depth known as the epicranial aponeurosis, also called the galea aponeurotica.

This retrospective study, examines the tumor- en surgical characteristics of these stage T3 cutaneous squamous cell carcinomas on the scalp.

ELIGIBILITY:
Inclusion Criteria:

* stage T3 cutaneous squamous cell carcinoma of the scalp (histologically proven)
* surgical treatment or radiotherapy treatment

Exclusion Criteria:

* metastasis by diagnosis
* stage T1/T2/T4

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Data from patients are collected retrospectively using data from the Pathological Anatomical National Automated Archive (PALGA) of the MUMC+ between 2010 - 2018. The TNM staging of all cutaneous squamous cell carcinomas in the research period was reassessed and classified following the TNM 8 criteria.
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2021-05-03 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Surgical characteristics | Between 2010-2017
  Choice of treatment, complications, reconstruction types
Tumor characteristics | Between 2010-2017
  Histological data on invasion depth, tumor differentiation
Patients characteristics | Between 2010-2017
  Risk factors, comorbidities

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Kelleners-Smeets, dr., Principal Investigator — Maastricht UMC
Locations (1):
- Ellen Oyen, Maastricht, Netherlands

REFERENCES:
- [Background] Amin MB, Greene FL, Edge SB, Compton CC, Gershenwald JE, Brookland RK, Meyer L, Gress DM, Byrd DR, Winchester DP. The Eighth Edition AJCC Cancer Staging Manual: Continuing to build a bridge from a population-based to a more "personalized" approach to cancer staging. CA Cancer J Clin. 2017 Mar;67(2):93-99. doi: 10.3322/caac.21388. Epub 2017 Jan 17. PMID 28094848